CLINICAL TRIAL: NCT07109895
Title: Effects of a Polyethene-Poron Custom Insole Combined With Transcutaneous Electrical Nerve Stimulation on Clinical Outcomes in Diabetic Foot Ulcers
Brief Title: Custom Insole With Transcutaneous Electrical Nerve Stimulation on Clinical Outcomes of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Custom Insole with TENS
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: Functional Disability; Diabetic Foot Ulcer; Transcutaneous Electrical Nerve Stimulation; Customized Insole; Pain; Dynamic Balance; Risk of Fall; Wound Size; Wound Depth; Diabetes
MeSH Terms: conditions — Diabetic Foot; Pain; Diabetes Mellitus | interventions — Transcutaneous Electric Nerve Stimulation; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a four-arm parallel-group interventional study designed to evaluate the effects of transcutaneous electrical nerve stimulation (TENS), custom insoles, and their combination in addition to standard care in patients with diabetic foot ulcers (DFUs). Participants will be randomly assigned to one of the following groups:
  Group 1: Standard care alone Group 2: TENS + standard care Group 3: Custom insole + standard care Group 4: TENS + custom insole + standard care
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be kept blinded of treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care Only (Other): Participants will receive standard care for diabetic foot ulcers.
  Interventions: Other: Standard Care Only
- Custom Insole + Standard Care (Experimental): Participants will receive a custom insole along with standard care.
  Interventions: Other: Custom Insole + Standard Care
- TENS + Custom Insole + Standard Care (Experimental): Participants will receive TENS therapy, a custom insole, and standard care.
  Interventions: Other: TENS + Custom Insole + Standard Care
- TENS + Standard Care (Experimental): Participants will receive transcutaneous electrical nerve stimulation (TENS) in addition to standard care.
  Interventions: Other: TENS plus Standard Care

INTERVENTIONS:
Other: Standard Care Only — Standard care includes routine wound debridement, moist wound dressings infection control, glycemic management, vascular assessment, and patient education in line with international DFU management guidelines.
  Arms: Standard Care Only
Other: TENS plus Standard Care — This experimental group will receive the same intervention plus Transcutaneous Electrical Nerve Stimulation (TENS) in burst mode (1-4 Hz at 100 Hz) applied around the wound site for 30 minutes, along with standard care.
  Arms: TENS + Standard Care
Other: Custom Insole + Standard Care — The experimental group will receive customised polyethene foam insoles with a Poron top layer along with standard care.
  Arms: Custom Insole + Standard Care
Other: TENS + Custom Insole + Standard Care — Participants in this group will receive a combination of transcutaneous electrical nerve stimulation (TENS), custom-made insole therapy, and standard care for diabetic foot ulcers (DFUs).
  Arms: TENS + Custom Insole + Standard Care

SUMMARY:
Diabetic foot ulcers (DFUs) are one of the serious complications of diabetes, typically resulting from neuropathy or peripheral arterial disease, and can often lead to amputation. It affects approximately 6.3% of people with diabetes globally. In Pakistan, the overall prevalence of DFUs is 16.83%, with a slightly higher rate in females. Diabetic foot ulcers are the main reason for lower extremity amputation (LEA) with non-traumatic origin, hospitalization, healthcare costs, and mortality.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) are a significant complication of diabetes, carry a high risk of amputation and disability, and affect around 6.3% of diabetic patients globally. Risk factors for DFUs include pre-ulcerative lesions, mechanical pressure, restricted mobility, and poor glycemic control. Peripheral neuropathy plays a crucial role in DFU development, causing structural and functional changes in the foot.

Offloading interventions, such as prefabricated orthotics and custom insoles, are essential for preventing DFU development and promoting ulcer healing. Physiotherapy modalities like therapeutic exercise and electrotherapy can assist in tissue repair and pain management. Orthotic management complements rehabilitation efforts, potentially reducing the risk of wound development. Further research on the combined benefits of transcutaneous electrical nerve stimulation (TENS) and customized insoles for DFUs is necessary to enhance clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old with type 1 and 2 diabetes
2. Both Males and Females
3. Having Foot ulcers in Grade 1 and Grade 2 according to the Wagner Classification

Exclusion Criteria:

1. History of amputation (proximal to the trans-metatarsal joint)
2. Active or inactive Charcot foot
3. Non-constructible peripheral vascular disease secondary to arteriosclerosis (AS)
4. Leg length discrepancy
5. The presence of any allergic condition of the skin,
6. Chronic consumption of opioids,
7. Use of a cardiac pacemaker,
8. Major bone operation,
9. Neurological illness, such as a vestibular disorder with a history of dizziness 10. Mental disorders, which might interfere with the assessment process

11. Dementia or impaired cognitive function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be measured at baseline, and change in pain intensity will be measured at 4th week, 8th week, and 12th week.
  Pain intensity will be measured using a visual analogue scale. It is an 11-point scale where "0" indicates no pain and "10" indicates the worst possible pain.
Dynamic Balance: | Change in status of dynamic balance will be measured at 4th week, at 8th week and 12th week of treatment.
  The time up and go (TUG) scale will be used for measuring dynamic balance. A time score of ≤10 seconds is considered normal, and a time of ≥14 seconds has been shown to indicate a high risk of falls.
Wound Healing | Wound dimensions will be measured at baseline, and change in length and width will be measured at the 4th week, 8th week, and 12th week of the treatment session.
  Patients will be assessed for ulcer dimensions by using a simple ruler method. Length and width will be noted using a simple ruler method.

SECONDARY OUTCOMES:
Risk of fall | Risk of fall will be measured at baseline, and change in status will be measured at the 4th week, 8th week, and 12th week of the treatment session.
  The Tinetti Scale will be used to measure the risk of fall. The final score of the scale is 28 points, and the interpretation is as follows: 25-28 = low risk of falls; 19-24 = moderate risk of falls; and <19 = high risk of falls.
Toe Muscle Strength | Toe Muscle Strength will be measured at baseline, and change in strength will be measured at the 4th week, 8th week, and 12th week of the treatment session.
  The paper grip test (PGT) will be used to measure toe muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ashfaq Ahmed, PhD Physiotherapy, Study Director — University of Lahore
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Will be share after publication